CLINICAL TRIAL: NCT06998472
Title: Evaluation of Pediatric Massage in the Treatment of Allergic Rhinitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Shu-Yu Yang, Director of the Department of Pediatrics, Division of Traditional Chinese Medicine, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 111-31
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Enhancing Treatment Outcomes for Patients With Allergic Rhinitis
Keywords: Tuina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Maintain the original treatment approach
  Interventions: Other: Maintain the original treatment approach
- tuina group (Experimental): Tuina therapy is administered once a week, each session lasting 15 minutes, for a duration of three months
  Interventions: Other: Tuina

INTERVENTIONS:
Other: Tuina — According to traditional Chinese medicine (TCM), children's physiological characteristics include immature and delicate internal organs, as well as underdeveloped qi and physical form. Pathologically, their organ systems are described as light and responsive, meaning they react quickly to both internal and external stimuli. Therefore, pediatric tuina must prioritize gentleness in technique. The applied pressure should not exceed 0.3 kilograms, and the depth of skin indentation should not go beyond 0.3 centimeters.
  Arms: tuina group
Other: Maintain the original treatment approach — Maintain the original treatment approach
  Arms: control group

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness of pediatric tuina (traditional Chinese pediatric massage therapy) in children with allergic rhinitis, aiming to provide an effective, non-invasive treatment option. This study will last for 12 weeks. If you meet the eligibility criteria, agree to participate, and sign the informed consent form, you will be randomly assigned to one of two groups: the treatment group or the control group. Random assignment is similar to a dice roll, giving you a 50% chance of being placed in either group.

Participants in the treatment group will receive pediatric tuina in combination with standard Western medical treatment. Participants in the control group will receive only the standard Western medical treatment. At the beginning of the trial, a pediatrician will collect your medical history and basic information. In addition, a traditional Chinese medicine (TCM) practitioner will conduct a meridian energy assessment and perform a TCM diagnostic evaluation (including the Four Diagnostic Methods and Heat Syndrome Assessment), which will take approximately 20 minutes. A research assistant will help administer a 22-item nasal symptom questionnaire and an allergic rhinitis quality of life questionnaire, which will take about 10 minutes. During the 12-week treatment period, follow-up assessments will be conducted twice-once at week 4 and again at the end of the treatment period in week 12. Both follow-ups will include the meridian energy test, TCM diagnostic evaluation, and allergic rhinitis questionnaires. Throughout the 12-week trial, participants in the treatment group will receive pediatric tuina therapy once a week. Each session will last approximately 15 minutes and will be conducted by a licensed TCM practitioner on a treatment table in the clinic.

The pediatric tuina treatment in this study will primarily focus on regulating the Bladder Meridian (dorsal fascia), Stomach Meridian (abdominal fascia), and the Lower Jiao (pelvic region). The techniques used are based on the Formless Qi Manipulation Tuina method developed by Master Chen Ming-Tang.

The treatment sequence begins with the "Swimming Belt to Search for Food" technique, which is used to relax the upper and middle segments of the spine, release tension in the paraspinal muscles, and correct spinal distortions. This is followed by the "Scooping Water to Splash the Face" technique to loosen the lower spine and pelvic region, helping to restore balance and alignment in the pelvis. Finally, the "Master Pulling the Spinning Top" technique is used to regulate the tibia, thereby improving gait and correcting imbalances in the pelvis and spine caused by improper walking posture.

The goal of this tuina treatment is to restore the body's structural balance. By adjusting muscles, tendons, ligaments, and fascia back to their proper alignment, qi and blood can circulate smoothly throughout the body. This supports the TCM principle that "when vital qi is strong, pathogenic factors cannot invade," thereby promoting a healthy internal environment.

The Meridian Energy Analysis Device (MEAD) is a computerized, non-invasive diagnostic tool commonly used in traditional Chinese medicine. It measures the activity level of the body's meridians and helps provide more accurate diagnostic insight from a TCM perspective. During the test, the practitioner will ask you to hold a testing probe while another probe touches 24 specific acupuncture points around the wrists and ankles. The assessment takes approximately 20 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* (1) no skin surface damage (2) no mental or cognitive impairments, with clear consciousness, and (3) a patient who has been medically diagnosed with allergic rhinitis.

Exclusion Criteria:

* (1) the presence of inflammatory wounds or ulcers on the skin surface; (2) pregnant or breastfeeding women; (3) individuals with congenital genetic diseases, heart disease, tumors, or chronic illnesses.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | This study will last for 12 weeks. During this 12-week trial period, participants will receive pediatric Tuina therapy once a week. A follow-up assessment will be conducted at Week 16. Eligibility
  The evaluation of allergic rhinitis symptom efficacy is measured using the RQLQ. The RQLQ consists of 28 questions across seven domains: activity limitations, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems, sleep problems, and emotional function Additionally, there are three patient-specific activity-related questions, allowing patients to select the three activities they most frequently engage in that are restricted by their allergic rhinitis symptoms. Subjects respond to each question using a 7-point scale (0 = not impaired at all, 6 = severely impaired). The overall RQLQ score is calculated as the mean of all 28 responses, while the domain scores represent the average score of items within each respective domain.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Yang, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taichung Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes